CLINICAL TRIAL: NCT04151329
Title: Evaluation for the Safety of BAT1306 and BAT8001 Injection for the Treatment of Patients With HER2-positive Advanced Solid Tumors Phase I/IIa Clinical Trials of Sexual, Tolerability and Pharmacokinetic Characteristics
Brief Title: A Phase I Clinical Trial of BAT1306 and BAT8001 Injection in Patients With Solid Tumor
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BAT-8001+1306-001GC-CR
Record Dates: First submitted 2019-10-30; First posted 2019-11-05 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-06

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2.4mg/kg of BAT8001 (Experimental): Drug:BAT1306 100mg/4ml/box, 200mg IV infusions ,BAT8001 100mg/box, 2.4mg/kg IV infusions
  Interventions: Biological: BAT1306 and BAT8001 2.4mg/kg
- 3.6mg/kg of BAT8001 (Experimental): Drug:BAT1306 100mg/4ml/box, 200mg IV infusions ,BAT8001 100mg/box,3.6mg/kg IV infusions
  Interventions: Biological: BAT1306 and BAT8001 3.6mg/kg

INTERVENTIONS:
Biological: BAT1306 and BAT8001 2.4mg/kg — Phase 1 dose titration study of BAT1306 and BAT8001 2.4mg/kg , then choose a proper dose for amplification study based on DLT result
  Arms: 2.4mg/kg of BAT8001
Biological: BAT1306 and BAT8001 3.6mg/kg — Phase 1 dose titration study of BAT1306 and BAT8001 3.6mg/kg , then choose a proper dose for amplification study based on DLT result
  Arms: 3.6mg/kg of BAT8001

SUMMARY:
A Phase I Clinical Trial of BAT1306 and BAT8001 Injection in Patients With HER2-positive Advanced Solid Tumor

DETAILED DESCRIPTION:
main purpose: To evaluate the safety and tolerability of BAT8001 in combination with BAT1306 in patients with HER2-positive advanced solid tumors, and to explore the maximum tolerated dose (MTD) to determine the recommended dose for phase II clinical trials (RP2D). Secondary purpose: (1) Evaluation of pharmacokinetic (PK) and immunogenic characteristics of BAT8001 in combination with BAT1306. (2) Preliminary evaluation of the antitumor efficacy of BAT8001 in combination with BAT1306. Exploratory purpose: To explore the efficacy-related biomarkers of BAT8001 in combination with BAT1306 in the treatment of patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 75 (inclusive) years old male and female;
2. Patients with advanced malignant solid tumors confirmed by histology or cytology, who have failed standard treatment, or who have no standard treatment plan, or who are not suitable for standard treatment at this stage;
3. Confirmed by the test as HER2 positive, defined as: IHC 3+ or ISH +;
4. ECOG physical status score 0-1 points;
5. Estimated survival time of more than 3 months;
6. According to RECIST version 1.1, there is at least one measurable tumor lesion;
7. Have adequate organ function: (1) Blood system (no blood transfusion or colony stimulating factor (G-CSF) treatment within 14 days): Neutrophil absolute value (ANC) ≥1.5×10^9/L; Platelet (PLT) ≥100×10^9/L; Hemoglobin (Hb) ≥90g/L; (2) liver function: Total bilirubin (TBIL) ≤1.5×ULN; Alanine aminotransferase (ALT) ≤ 2.5 × ULN; Aspartate aminotransferase (AST) ≤ 2.5 × ULN; (3) Renal function: Creatinine (Cr) ≤ 1.5 × ULN; Creatinine clearance (CCr) >50ml/min (calculated according to Cockcroft-Gault formula); Coagulation; Activated partial thromboplastin time (APTT) ≤ 1.5 × ULN; International normalized ratio (INR) ≤ 1.5 × ULN; Myocardial zymogram; Troponin T <1×ULN;
8. Qualified patients (male and female) with fertility must agree to use reliable methods of contraception (hormone or barrier or abstinence) during the trial period and at least 6 months after the last dose; female patients of childbearing age are selected before the election. The blood pregnancy test within the day must be negative;
9. Subjects must give informed consent to the study prior to the trial and voluntarily sign a written informed consent form.

Exclusion Criteria:

1. Receive anti-tumor therapy such as radiotherapy, chemotherapy, targeted therapy, endocrine therapy or immunotherapy within 4 weeks before the first dose, or other clinical trial drug treatment; Note: Immunological checkpoint inhibitors, including anti-PD-1 antibody, anti-PD-L1 antibody, mitomycin and nitrosourea for 6 weeks from the last dose; fluorouracil oral drugs such as tegao, card Peitabin is within 2 weeks of taking the last dose; 2. The cumulative dose of anthracycline used in the past meets any of the following values: Doxorubicin or liposomal doxorubicin >360mg/m2 ? Epirubicin > 540mg/m2 ? Mitoxantrone > 84mg/m2
2. If another anthracycline or more than one anthracycline is used, the cumulative dose exceeds the equivalent dose of doxorubicin 360 mg/m2
3. Have undergone major organ surgery (excluding needle biopsy) or significant trauma within 4 weeks prior to the first dose; subcutaneous venous access device implantation (eg PICC) within 7 days;
4. Need to be combined during the trial, or 1 week before the first dose (or 3 half-lives of the drug, whichever is longer), have received strong inducers or strong inhibitors of CYP3A4 (see Appendix 7);
5. Adverse reactions to previous anti-tumor treatment have not been restored to CTCAE 5.0 grade evaluation ≤ 1 (except for hair loss);
6. Brain metastases with clinical symptoms, spinal cord compression, cancerous meningitis, or other evidence that the central nervous system metastases in patients have not been controlled, the researchers judged that it is not suitable for enrollment; patients with clinical symptoms suspected of brain or pia mater Need to be excluded by CT / MRI examination; 7.
7. There have been ≥3 immune-related adverse events (irAE, see Appendix 5) in immunotherapy.
8. Patients with active or pre-existing autoimmune diseases that may have recurrence (eg, systemic lupus erythematosus, rheumatoid arthritis, vasculitis, etc.); 9. Patients who have received systemic corticosteroids (prednisone >10 mg/day or equivalent dose of the same drug) or other immunosuppressive agents within 14 days prior to the first dose; Except for the use of topical, ocular, intra-articular, intranasal, and inhaled corticosteroids; short-term use of corticosteroids for prophylaxis, such as the use of contrast agents;

10. Currently or have had interstitial lung disease; 11. There are uncontrolled active infections; 12. Have a history of immunodeficiency, including HIV antibody test positive; 13. Active hepatitis B patients (hepatitis B virus titer is higher than the lower limit of detection), allowing prophylactic antiviral therapy other than interferon; hepatitis C virus infection (anti-hepatitis C antibody positive or hepatitis C RNA) Positive); 14. There are ≥2 grade peripheral neuropathy; 15. Have a history of serious cardiovascular disease: ? Ventricular arrhythmias requiring clinical intervention; Acute coronary syndrome, congestive heart failure, stroke, thromboembolic events, or other cardiovascular events of grade 3 or above within 6 months prior to enrollment; 15.New York Heart Association (NYHA) cardiac function classification ≥ II or left ventricular ejection fraction (LVEF) < 50%; 16. Hypertension that cannot be controlled by a single drug (systolic blood pressure after treatment >140 mmHg and/or diastolic blood pressure >90 mmHg); 16. Known to be allergic to trastuzumab or other anti-PD-1, anti-PD-L1 monoclonal antibody drugs; 17. Alcohol or drug dependence is known; 18. Persons with mental disorders or poor compliance; 19. Women during pregnancy or lactation; 20. The investigator believes that the subject has any clinical or laboratory abnormalities or other reasons that are not suitable for participation in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2019-06-21 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity（DLT） | 3weeks
  Safety and tolerability endpoint
Area under the curve (AUC) | 3weeks
  Pharmacokinetic endpoint
Maximum serum drug concentration (Cmax) | 3weeks
  Pharmacokinetic endpoint
Half-life period(t1/2) | 3weeks
  Pharmacokinetic endpoint
Anti drug antibodies (ADA) | through study completion, an average between half year and a year
  Plasma level of anti drug antibodies (ADA) correlated with bevacizumab plasma level
Neutralizing anti-drug antibodies (NADA) | through study completion, an average between half year and a year
  Neutralizing anti-drug antibodies (NADA) correlated with bevacizumab plasma level

SECONDARY OUTCOMES:
ORR | through study completion, an average between half year and a year
  Overall response rate
PFS | through study completion, an average between half year and a year
  Progression free survival time
DCR | through study completion, an average between half year and a year
  Disease control rate
DOR | through study completion, an average between half year and a year
  Duration of response

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Ethics Committee of Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Undecided